CLINICAL TRIAL: NCT07323875
Title: Single-Row Versus Double-Row Repair in the Surgical Management of Achilles Insertional Tendinopathy: A Randomized Controlled Trial (STRIDE Trial)
Brief Title: Single-Row Versus Double-Row Repair for Achilles Insertional Tendinopathy
Acronym: STRIDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); University Health Network, Toronto (Other); Unity Health Toronto (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Sam Park, MD MASc FRCPC, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTO Study Number:5686
Record Dates: First submitted 2025-11-28; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Achilles Insertional Tendinopathy; Achilles Tendinopathy
Keywords: single row repair; double row repair; calcaneal insertion

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized controlled clinical trial of patients undergoing surgical management for chronic Achilles insertional tendinopathy.
Who Masked: Participant, Outcomes Assessor
Masking Description: As noted above, only the surgeon will be aware of allocation assignment. The participant and outcomes assessors will be blinded to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-row repair Arm (Active Comparator): Single-row repair will involve 2 suture anchors (2 anchors total)
  Interventions: Procedure: Single-row repair of the Achilles tendon at its calcaneal insertion
- Double-row repair Arm (Active Comparator): Double-row repair will involve 2 suture anchors for the proximal row and 2 suture anchors for the distal row (4 anchors total)
  Interventions: Procedure: Double-row repair of the Achilles tendon at its calcaneal insertion

INTERVENTIONS:
Procedure: Single-row repair of the Achilles tendon at its calcaneal insertion — single-row (2 anchors)
  Arms: Single-row repair Arm
Procedure: Double-row repair of the Achilles tendon at its calcaneal insertion — double-row (4 anchors)
  Arms: Double-row repair Arm

SUMMARY:
Achilles insertional tendinopathy may require surgical debridement and tendon reattachment when non-operative treatment fails. Single-row and double-row repairs are used, with biomechanical studies favoring double-row, but clinical evidence of improved outcomes is lacking and costs are higher. This multi-center randomized trial will use the VISA-A score to compare outcomes and inform cost-effective, evidence-based surgical care.

DETAILED DESCRIPTION:
Double-row repairs for Achilles insertional tendinopathy have been shown biomechanically to be stronger than single-row repairs, but clinical studies have not demonstrated clear advantages. Existing comparative studies are limited by retrospective designs and use of non-validated outcome measures such as AOFAS, VAS, and SF-36 Physical Function. No prospective randomized trials have evaluated clinical outcomes of single-row versus double-row repairs.

This multi-center randomized controlled trial will use the disease-specific Victorian Institute of Sports Assessment-Achilles (VISA-A) score to compare clinical outcomes between single-row and double-row repairs, providing high-quality evidence to guide optimal surgical management.

ELIGIBILITY:
Inclusion Criteria:

1. Must be deemed to have capacity to provide informed consent;
2. Must sign and date the informed consent form;
3. Stated willingness to comply with all study procedures;
4. Adult patients between the ages of 18 and 75 years with symptomatic chronic Achilles insertional tendinopathy for a minimum of 3 months
5. Failure of non-operative management (which includes physiotherapy, stretching exercises, heel lifts, nonsteroidal anti-inflammatory drugs (NSAIDs), activity modification, etc.) for at least 3 months.
6. Preoperative imaging (x-ray and Medical Resonance Imaging (MRI)) is available and completed;
7. Willingness of patients to follow the postoperative rehabilitation protocol;
8. Willingness of patients to be available for follow up appointments for up to 2 years.

Exclusion Criteria:

1. Non-insertional Achilles tendinopathy;
2. Achilles tendon rupture;
3. Previous Achilles tendon surgery;
4. Oral steroid use or steroid injection within 3 months of surgery;
5. History of connective tissue or collagen disorder (e.g. Marfan Syndrome)
6. History of chronic inflammatory disorders
7. History of neurological disease (stroke, cerebral palsy)
8. History of using more than 30mg of oxycodone or equivalent per day;
9. Current cigarette smoker (Former smokers must have quit for minimum of one year)
10. Diabetes type I or II
11. Pregnancy
12. Hypersensitivity to metal, Polylactic Acid (PLA), or Polyetheretherketone (PEEK) materials
13. Active infection
14. Worker's compensation claim (e.g. WSIB)
15. History of cognitive or mental health conditions that would make the participant unable to complete study procedures
16. Non-English speaking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Disease-specific outcomes | 24 months after surgery
  The Victorian Institute of Sport Assessment-Achilles (VISA-A) questionnaire is a validated, self-reported outcome measure designed to assess the severity of Achilles tendinopathy. It evaluates three key domains: pain, function, and activity level and produces a score from 0 to 100, with higher scores indicating better function and fewer symptoms.

SECONDARY OUTCOMES:
Surgical Cost | Within 2 hours of surgery
  Assess the cost difference between single-row repair versus double-row repair
Foot and Ankle Ability Measure (FAAM) | 24 months after surgery
  The FAAM is a patient-reported outcome questionnaire designed to assess physical function in individuals with foot and ankle disorders.
  Scores are typically expressed as percentages, with higher scores indicating better function.
Visual Analogue Scale Foot and ankle (VAS-FA) | 24 months after surgery
  The VAS-FA is a patient-reported outcome measure designed to assess pain, function, and other symptoms related to foot and ankle disorders. It uses a visual analogue scale, typically a 100 mm line, where patients indicate the severity of their symptoms. Higher scores usually indicate better function or less pain.
Plantarflexion strength | 24 months after surgery
  Measured using a HUMAC Norm Isokinetic Dynamometer Weakness: May indicate calf muscle atrophy, nerve injury, or Achilles tendon dysfunction.
  Deficits: Can cause altered gait, decreased push-off, and balance problems.
Biomechanical performance | 24 months after surgery
  Including ankle kinematics and kinetics during gait and functional tasks, assessed through markerless motion tracking.
  Gait Analysis: Evaluating walking or running patterns in patients with musculoskeletal or neurological impairments.
Functional endurance | 24 months after surgery
  As measured by the Heel Rise Test
  Normal: Able to perform ≥25-30 single-leg heel raises with minimal fatigue. Weakness: Fewer repetitions or lower heel height may suggest calf muscle weakness.
Surgical Time | During surgery
  Assess the operative time required for single-row repair versus double-row repair.

CONTACTS AND LOCATIONS:
Overall Officials: Si-Hyeong Sam Park, MD, FRCPC, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada